CLINICAL TRIAL: NCT03273725
Title: The TRIP-Tooth Study: Maternal Pre- and Postnatal Vitamin D Levels and Dental Caries in Children 7-9 Years of Age.
Brief Title: Maternal Vitamin D Levels in Pregnancy and Dental Caries in Children
Status: Completed | Type: Observational
Sponsor: Tannhelsetjenestens Kompetansesenter Midt-Norge (Other)
Responsible Party: Principal Investigator, Tone Natland Fagerhaug, Head of Research, Tannhelsetjenestens Kompetansesenter Midt-Norge
Other Study IDs: TannhelsetjenestensKM
Record Dates: First submitted 2016-01-24; First posted 2017-09-06 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Vitamin D Deficiency; Dental Caries; Dental Enamel Hypoplasia
Keywords: Oral Health; Vitamin D
MeSH Terms: conditions — Vitamin D Deficiency; Dental Caries; Dental Enamel Hypoplasia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva samples
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Dental examination including taking a saliva sample. — The main focus of the dental examination is enamel defects and caries. Saliva samples (stimulated) will also be taken.

SUMMARY:
The main aim of this study is to investigate potential associations between maternal pre- and postnatal vitamin D level and oral health outcomes (caries and developmental defects of enamel) in their children at 7-9 years of age.

DETAILED DESCRIPTION:
Vitamin D plays an important part in calcium absorption needed for calcification of hard tissues such as bone. Lack of vitamin D can lead to growth retardation in children and a variety of bone related problems in adulthood such as osteopenia, osteoporosis and increased risk of bone fracture. Vitamin D deficiency has also been associated with a variety of other health problems. In relation to oral health, studies have suggested that lack of vitamin D may interfere with tooth development resulting in development defects of the enamel, which in turn increase the risk of dental caries. As teeth begin to calcify around 14 weeks in utero and continue until the enamel on the last primary tooth is completed around ten months after birth, it is plausible that both pre- and postnatal vitamin D levels can have an impact on the development of the enamel in primary teeth in the offspring, which in turn may be related to the risk of developing enamel defects and dental caries. Furthermore, vitamin D may play a role in the immune system and thereby affect the oral microflora. Vitamin D could therefore also affect the risk of caries through immunological pathways. Few previous studies have investigated the associations between vitamin D and oral health outcomes, such as these.

The aim of this study is to investigate the potential associations between maternal pre- and postnatal vitamin D levels and oral health outcomes, such as caries and dental enamel defects in the offspring at 7-9 years of age.

The current study is a follow-up study of a previous study conducted in Trondheim and Stavanger, Norway. In 2007-2009 a total of 855 pregnant women participated in the Training in Pregnancy (TRIP) study, a randomised controlled trial study conducted to investigate whether exercise during pregnancy would help prevent or treat various pregnancy related illnesses. The women were included between weeks 18-22 of pregnancy and were followed-up at week 32-36 of pregnancy and at 3 months post-partum. An additional follow-up was also conducted among the participants from Trondheim at 18 months post-partum. The data collection included both questionnaires, clinical examinations and blood samples. The blood samples taken from the mothers at 18-22 weeks and 32-36 weeks of pregnancy have been analysed for levels of vitamin D, calcium, phosphate, magnesium, creatinine, albumin and PTH. In the current study, the children are invited to a dental examination, including a saliva sample. These clinical examinations will be conducted from June 2016 through to August 2017.

ELIGIBILITY:
Inclusion Criteria:

* Mother of the child participated in the main study "Training in Pregnancy"

Exclusion Criteria:

* Consent not given

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All n=855 mother/child pairs who participated in the initial TRIP study in 2007-2009 will be invited to participate in the follow-up study in 2016-2017.
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Dental caries in the primary teeth of the children at the age of 7-9 yrs | 2016 - 2017
  The main study was conducted in 2007 - 2009. In the current study the children of the mothers participating in the main study are invited to the follow-up study "Trip Tooth Study" with data collection (dental examination) taking place over a time span of two years.

SECONDARY OUTCOMES:
Enamel defects in the primary teeth of the children at the age of 7-9 yrs | 2016 - 2017
  The main study was conducted in 2007 - 2009. In the current study the children of the mothers participating in the main study are invited to the follow-up study "Trip Tooth Study" with data collection (dental examination) taking place over a time span of two years.
Antimicrobial peptides in saliva | 2016 - 2017
  The main study was conducted in 2007 - 2009. In the current study the children of the mothers participating in the main study are invited to the follow-up study "Trip Tooth Study" with data collection (dental examination including a saliva sample) taking place over a time span of two years.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available for sharing data.